CLINICAL TRIAL: NCT05768971
Title: Conventional Ultrasound and Quantitative Dynamic Contrast-Enhanced Ultrasound (DCE-US) of the Bowel Wall in Patients With Food Allergy in Comparison to Crohn´s Disease and Healthy Controls
Brief Title: Contrast-enhanced Ultrasound in Patients With Crohn´s Disease and Food Allergy
Status: Completed | Type: Observational
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Dane Wildner, Principal Investigator - Deputy Head of Ultrasound Department, Department of Internal Medicine 1, Universitätsklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg
Other Study IDs: DCEUS_CD_NMA
Record Dates: First submitted 2023-02-28; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Crohn Disease; Food Allergy
MeSH Terms: conditions — Crohn Disease; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active Crohn´s disease: Ultrasound in patients with proven active Crohn´s disease scheduled for therapy with anti tumor necrosis factor alpha antibodies
- Patients with Food allergy: Patients with proven food allergy
  Interventions: Other: Mild diet; Other: Provocative diet
- Healthy controls: Healthy, food-tolerant volunteers without any abdominal complaint
  Interventions: Other: Mild diet; Other: Provocative diet

INTERVENTIONS:
Other: Mild diet
  Groups: Healthy controls; Patients with Food allergy
Other: Provocative diet
  Groups: Healthy controls; Patients with Food allergy

SUMMARY:
The purpose of this study is to investigate differences of the bowel wall thickness visible in conventional ultrasound and bowel perfusion using quantitative Contrast-Enhanced Ultrasound in patients with Crohn´s disease in comparison with healthy controls and patients with food allergy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written consent will undergo conventional transabdominal ultrasound and Contrast-Enhanced Ultrasound of the bowel wall with measurement of the bowel wall thickness. In addition a continuous video sequence during Contrast-Enhanced Ultrasound is recorded and perfusion kinetics from the video clips are analyzed using a specific quantification software.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Endoscopically and histologically confirmed active Crohn´s disease or
* Previously proven food allergy (double-blind or single-blind food challenge tests with placebo controls previously before the sonographic examination, increased blood and / or intestinal Immunoglobulin E levels, elevated methylhistamine values under provocation and with reproducible reactions during food challenge procedures) or
* Healthy individuals without abdominal complaints

Exclusion Criteria:

* Age under 18
* Intolerance of the ultrasound contrast agent SonoVue
* Refusal of participation in the study
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary-care university hospital, patients diagnosed and treated in the outpatient department for inflammatory and allergic bowel diseases
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2014-11-14 (Actual); Study Completion 2014-11-14 (Actual)

PRIMARY OUTCOMES:
Bowel wall thickness | T0: Baseline after mild diet. T1: After provocative diet (up to 30 days from T0)
  Thickness of the bowel wall measured in high-frequency ultrasound from the center of the lumen to the serosa
Peak Enhancement | T0: Baseline after mild diet. T1: After provocative diet (up to 30 days from T0)
  Maximum point of the DCE-US curve assessed in Contrast-Enhanced Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Dane Wildner, M.D., Principal Investigator — Department of Medicine 1, Divison of ultrasound medicine, University Hospital Erlangen

IPD SHARING:
Plan to Share IPD: No